CLINICAL TRIAL: NCT03096119
Title: A Study to Define the Distribution of Type of Hypertension in Asia by Blood Pressure Monitoring at Home (Asia BP@Home)
Acronym: Asia BP@Home
Status: Completed | Type: Observational
Sponsor: Jichi Medical University (Other)
Responsible Party: Principal Investigator, Kazuomi Kario, Professor & Chairman, Jichi Medical University
Other Study IDs: RinA16-080
Record Dates: First submitted 2017-03-23; First posted 2017-03-30 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Hypertension
Keywords: blood pressure monitoring, home; Asia
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: home blood pressure measurement — We ask participants to measure their home blood pressure 7 days or more.

SUMMARY:
Blood pressure variability (BPV) is being increasingly recognized as an important influence on hypertension outcomes as well as a risk factor for other cardiovascular (CV) events. However, in Asia there is a current lack of awareness of BPV and its significance on patient outcomes. Furthermore, there is ongoing debate on the role of home blood pressure (HBP) monitoring in managing hypertension patients and uncertainty on how best to integrate it into clinical practice.

Therefore, we conduct Asia BP@Home study to assess HBP control status in each Asian country and develop an Asian consensus and Asia-specific treatment for hypertension.

DETAILED DESCRIPTION:
Blood pressure variability (BPV) is being increasingly recognized as an important influence on hypertension outcomes as well as a risk factor for other cardiovascular (CV) events. However, in Asia there is a current lack of awareness of BPV and its significance on patient outcomes. Furthermore, there is ongoing debate on the role of home blood pressure (HBP) monitoring in managing hypertension patients and uncertainty on how best to integrate it into clinical practice.

The main purpose of this study is to:

* Assess HBP control status in each Asian country
* Develop an Asian consensus and Asia-specific treatment for hypertension
* Improve the management of hypertension in Asia by encouraging patients to monitor HBP

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 20 years
2. Subjects with stable medication (> 3 months) diagnosed as hypertension
3. Asian
4. Subjects have been thoroughly informed about this registry and signed an Informed Consent Form.

Exclusion Criteria:

-

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion criteria:
  1. Age >= 20 years
  2. Subjects with stable medication (> 3 months) diagnosed as hypertension
  3. Asian
  4. Subjects have been thoroughly informed about this registry and signed an Informed Consent Form.
Sampling Method: Non-Probability Sample
Enrollment: 1462 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Distribution rate based on the home BP of the patients. | 7 days or more blood pressure measurement
  Distribution rate based on the home BP of the patients who are defined as:
  * Masked morning hypertension
  * White-coat hypertension
  * Poorly controlled hypertension
  * Well controlled hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Kazuomi Kario, MD, PhD, Principal Investigator — Jichi Medical University School of Medicine
Locations (1):
- Jichi Medical University, Tochigi, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chia YC, Kario K, Tomitani N, Park S, Shin J, Turana Y, Tay JC, Buranakitjaroen P, Chen CH, Hoshide S, Nailes J, Minh HV, Siddique S, Sison J, Soenarta AA, Sogunuru GP, Sukonthasarn A, Teo BW, Verma N, Zhang Y, Wang TD, Wang JG. Comparison of day-to-day blood pressure variability in hypertensive patients with type 2 diabetes mellitus to those without diabetes: Asia BP@Home Study. J Clin Hypertens (Greenwich). 2020 Mar;22(3):407-414. doi: 10.1111/jch.13731. Epub 2019 Dec 31. PMID 31891447